CLINICAL TRIAL: NCT06682897
Title: Simplified Tai Chi Exercises to Improve Function in People With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Qian Qian, Principal Investigator, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17526
Record Dates: First submitted 2024-10-28; First posted 2024-11-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Chronic Ankle Instability
Keywords: ankle; Tai Chi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants will be asked to choose three time slots per week to come to the lab, and each time slot will consist of a 1-hour workout that includes a 10-minute warm-up, a 45-minute Tai Chi practice, and a 5-minute cool-down.
  Interventions: Behavioral: Tai Chi training
- Control (No Intervention): Participants replicated all the procedures of the exercise trial except for the different starting phase of the training.

INTERVENTIONS:
Behavioral: Tai Chi training — 60 minutes each session, three sessions per week, lasting 4 weeks for undertaking.
  Arms: Exercise

SUMMARY:
The goal of this interventional trial is to evaluate the effectiveness of the simplified four-week Tai Chi training in improving function in people with chronic ankle instability. The main questions it aims to answer are:

1. Does the 4-week Tai Chi training improve ankle neuromuscular responses?
2. Does the 4-week Tai Chi training enhance ankle proprioception?
3. Does the 4-week Tai Chi training improve ankle muscle strength？
4. Does the 4-week Tai Chi training boost balance performance？
5. Does the 4-week Tai Chi training enhance subjective ankle stability and quality of life?

Researchers will compare Tai Chi training to self-management to see if this Tai Chi training works to enhance ankle stability performance.

Participants will:

1. Take self-management and Tai Chi training, and each for 4 weeks
2. Visit the labs every 4 weeks for biomechanical measurements and questionnaires, totally 3 times.

DETAILED DESCRIPTION:
Tai Chi is a traditional Chinese exercise practiced by millions worldwide to stay active and improve health. Based on muscle activation levels across the full set of movements (108 forms), we developed a simplified 16-form Tai Chi routine to enhance ankle stability for individuals with chronic ankle instability.

To evaluate the benefits of this simplified 16-form version for ankle function in people with chronic ankle instability, we are recruiting individuals managing symptoms of chronic ankle instability for a 4-week training program and assess their ankle-related function three times. All participants are randomly allocated to both the Tai Chi training group or a self-management control group, while maintaining their usual lifestyle and exercise routines throughout the study. All participants will complete the same training content and assessment tasks; participants in the control group will be offered the Tai Chi training following completion of the second outcome assessment.

The Tai Chi training includes a total of 12 sessions over 4 weeks, with three sessions per week, each lasting 1 hour (10 minutes of warm-up, 45 minutes of Tai Chi practice, and a 5-minute cool down). Each of the three functional assessments will include consistent measures, including muscle activation, proprioception, muscle strength, balance testing, and self-assessment scales (ankle function and quality of life).

ELIGIBILITY:
Inclusion criteria:

* Aged from 18 to 40
* A history of at least one significant lateral ankle sprain was associated with inflammatory symptoms (pain, swelling, etc) and disrupted activity
* The initial sprain must have occurred at least 12 months prior to study enrolment
* The most recent injury must have occurred more than 3 months prior to study enrolment
* Reports of feeling instable or "giving way" during daily activities or physical activities and experienced at least 2 episodes in the 6 months prior to study enrolment
* Scoring ≤25 on the Cumberland Ankle Instability Tool

Exclusion criteria:

* Any previous fractures or surgeries on the lower limbs
* Have other muscle, joint or nerve disorders that affect the function of the lower limbs
* Chest pain at rest, dizziness during rest, heart condition, or doctor's advice not to exercise without medical supervision
* Currently enrolled in other ankle rehabilitation programmes
* Already a Tai Chi practitioner
* Pregnant
* Allergic to adhesive tapes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Ankle neuromuscular reponses | From the date of randomization until the completion of three assessments. This evaluation will be conducted at 0, 4, and 8 weeks after enrollment, with a maximum duration of 8 weeks.
  This includes two tasks, one is drop-landing, the other is ankle inversion perturbation. Each side will perform each task three times. Six electromyography muscle sensors will be placed on peroneus longus, peroneus brevis and tibialis anterior muscles to record muscle activity.

SECONDARY OUTCOMES:
Ankle proprioception | From the date of randomization until the completion of three assessments. This evaluation will be conducted at 0, 4, and 8 weeks after enrollment, with a maximum duration of 8 weeks.
  Proprioception will be tested using both the Humac Norm dynamometer and the trapdoor devices.
  Humac: Participants' ankles will be moved to inversion positions of 10 and 20 degrees and eversion positions of 10 and 15 degrees under the Humac device. The degrees of their active and passive replication will be recorded.
  Trapdoor: The tilt angle will be adjusted using four wooden blocks to 10, 12, 14, and 16 degrees. Each angle will be repeated randomly 10 times, totaling 40 trials. The perceived height number for each trial will be recorded.
Ankle muscle strength | From the date of randomization until the completion of three assessments. This evaluation will be conducted at 0, 4, and 8 weeks after enrollment, with a maximum duration of 8 weeks.
  Ankle Muscle Strength will be assessed using the HUMAC Norm dynamometer. The assessment of eversion will be conducted at a speed of 30°/s (eccentric and concentric), and inversion will be conducted at a speed of 60°/s (eccentric and concentric). The peak of the participant's maximum effort three times will be recorded.
Balance performance | From the date of randomization until the completion of three assessments. This evaluation will be conducted at 0, 4, and 8 weeks after enrollment, with a maximum duration of 8 weeks.
  Static balance:
  Participants are asked to complete three trials of unipedal stance on both limbs in both open and close eyes. A total of 12 trials are required, with each trial lasting for 10 s.
  Dynamic balance:
  SEBT: Three times each side. The most distal aspect of the great toe on 0 (crossroad of eight lines) during the entire procedure.The maximum distance (centimeters) for each reach direction is recorded.
  DLBT: Three times each side. All participants start by moving their right leg clockwise and their left leg counterclockwise to each direction. After jumping to an outer target, participants need to return to the center target and stabilise for two seconds, then jump again to an outer target. The total time will be recorded.
Questionnaire | From the date of randomization until the completion of three assessments. This evaluation will be conducted at 0, 4, and 8 weeks after enrollment, with a maximum duration of 8 weeks.
  This includes the assessment of subjective ankle stability using the Cumberland Ankle Instability Tool and the Foot and Ankle Ability Measure questionnaire, as well as the evaluation of quality of life using the SF-12 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional data protection policies.